CLINICAL TRIAL: NCT01043887
Title: A Single Dose Study to Investigate the Pharmacokinetics of Ridaforolimus in Patients With Hepatic Insufficiency
Brief Title: Ridaforolimus in Patients With Hepatic Insufficiency (MK-8669-046)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8669-046; MK8669-046; 2009_706
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Healthy Volunteers; Hepatic Insufficiency
Keywords: Healthy Volunteers; Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with Moderate Hepatic Insufficiency (Experimental): Patients with moderate hepatic insufficiency (a score of 7 to 9 on the Child-Pugh's scale) received a single 10 mg dose of ridaforolimus.
  Interventions: Drug: ridaforolimus
- Healthy Control Subjects (Experimental): Healthy control subjects were matched by race, age, gender, and body mass index (BMI) to the patients with moderate hepatic insufficiency. The healthy control subjects also received a single 10 mg dose of ridaforolimus.
  Interventions: Drug: ridaforolimus

INTERVENTIONS:
Drug: ridaforolimus — single oral dose administration 10 mg ridaforolimus

SUMMARY:
This study will evaluate the pharmacokinetics of ridaforolimus including the area under the concentration-time curve (AUC[0-infinity]) and maximum concentration (Cmax) after administration of a single dose of ridaforolimus in patients with moderate hepatic insufficiency and healthy matched control subjects.

ELIGIBILITY:
Inclusion Criteria:

Hepatic Patients:

* Female patient is of non-child bearing potential
* Apart from hepatic insufficiency with features of cirrhosis, patient is otherwise in good health
* Patient has a diagnosis of chronic stable hepatic insufficiency with features of cirrhosis

Healthy Subjects:

* Female subject is of non-childbearing potential
* Subject is in good health

Exclusion Criteria:

Hepatic Patients and Healthy Subjects:

* Works a night shift and is not able to avoid night shift work during the study
* Has a history of stroke, seizure or major neurological disease
* Has a history of cancer
* Is unable to refrain from or anticipates the use of any prescription or non-prescription drugs during the study
* Consumes excessive amounts of alcohol or caffeine
* Has had major surgery, donated blood or participated in another investigational study in the past 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC[0-infinity]) of ridaforolimus following a single oral dose. | 288 hours postdose
Maximum Concentration (Cmax) of ridaforolimus following a single oral dose. | 288 hours postdose
Tmax of a Single Oral Dose of Ridaforolimus. | 288 hours postdose
Apparent Terminal Half-life (t1/2) of a Single Oral Dose of Ridaforolimus. | 288 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC